CLINICAL TRIAL: NCT04704843
Title: A Phase 1b, Randomized, Double-Blind, Placebo-Controlled Study to Assess the Safety, Pharmacokinetics, Pharmacodynamics and Clinical Response of Guselkumab in Adult Participants With Celiac Disease
Brief Title: A Study of Guselkumab in Adult Participants With Celiac Disease
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Study terminated. Sponsor decision.
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR108914; 2020-003539-40 (EudraCT Number); 64304500CLD1001 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2021-01-08; First posted 2021-01-12 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Celiac Disease
MeSH Terms: conditions — Celiac Disease | interventions — guselkumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Module A (Without Gluten-Challenge): Guselkumab or Placebo (Experimental): Participants in Module A (without gluten-challenge) will receive intravenous (IV) infusion of guselkumab or matching placebo as induction dose at every 4 weeks through Week 8 followed by subcutaneous (SC) injection of guselkumab or matching placebo at Week 12.
  Interventions: Drug: Guselkumab; Drug: Placebo
- Module B (With Gluten-Challenge): Guselkumab or Placebo (Experimental): Participants in Module B (with gluten-challenge) will receive IV infusion of guselkumab or matching placebo as induction dose at every 4 weeks through Week 8 followed by SC injection of guselkumab or matching placebo at Week 12.
  Interventions: Drug: Guselkumab; Drug: Placebo

INTERVENTIONS:
Drug: Guselkumab — Guselkumab will be administered as IV infusion (induction dose) and SC injection.
Drug: Placebo — Matching placebo to guselkumab will be administered as IV infusion (induction dose) and SC injection.

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of guselkumab compared to placebo in participants with celiac disease.

ELIGIBILITY:
Inclusion Criteria:

* Have a body mass index (BMI) 16 to 45 kilogram per meter square (kg/m^2). Underweight participants (BMI 16 to 18 kg/m^2) may only be included if in the opinion of the investigator a participant was underweight due to active celiac disease and thus, may benefit from therapy but yet not be at significantly increased risk due to severe malabsorption or other conditions
* Physician-diagnosed celiac disease with documented history of biopsy-proven celiac disease
* Self-reported to be on a gluten-free diet (GFD) for at least 11 consecutive months prior to enrollment and have the willingness to continue to adhere to the same GFD while on study
* Willing to take/ingest gluten-containing product at specific study timepoints only (if assigned to Module B)
* Willing to undergo up to 3 on-study esophagogastroduodenoscopy (EGD) with biopsies

Exclusion Criteria:

* Has a history of chronic inflammatory gastrointestinal disease (example, inflammatory bowel disease, extensive colitis, ulcerative jejunitis, eosinophilic esophagitis)
* Has chronic infectious gastrointestinal illness, or acute infectious gastrointestinal illness within the 4-week period prior to screening
* Currently has a malignancy or a history of malignancy within 5 years before screening (with the exception of a non-melanoma skin cancer that has been adequately treated with no evidence of recurrence for at least 3 months before the first study intervention administration or cervical carcinoma in situ that has been treated with no evidence of recurrence for at least 3 months before the first study intervention); known history of lymphoproliferative disease, including monoclonal gammopathy of unknown significance, lymphoma, or signs and symptoms suggestive of possible lymphoproliferative disease, such as lymphadenopathy and/or splenomegaly
* Has a history of, or ongoing, chronic or recurrent infectious disease, including but not limited to, chronic renal infection, chronic chest infection, recurrent urinary tract infection (example, recurrent pyelonephritis or chronic non-remitting cystitis), or open, draining, or infected skin wounds or ulcers
* Has had previous treatment with guselkumab

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-06-17 (Actual); Primary Completion 2021-09-13 (Actual); Study Completion 2021-09-13 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Treatment-emergent Adverse Events (TEAEs) | Up to Week 28
  An adverse event (AE) is any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/biological agent under study. TEAEs are AEs with onset during the treatment phase or that are a consequence of a pre-existing condition that has worsened since baseline.
Number of Participants with Treatment-emergent Serious Adverse Events (SAEs) | Up to Week 28
  TEAEs are AEs with onset during the treatment phase or that are a consequence of a pre-existing condition that has worsened since baseline. A SAE is any untoward medical occurrence that at any dose: results in death; is life-threatening; requires inpatient hospitalization or prolongation of existing hospitalization; results in persistent or significant disability/incapacity; is a congenital anomaly/birth defect; is a suspected transmission of any infectious agent via a medicinal product; is medically important.
Number of Participants with Clinically Significant Abnormalities in Vital Signs | Up to Week 28
  Number of participants with clinically significant vital signs abnormalities including temperature, pulse/heart rate, respiratory rate, and blood pressure (systolic and diastolic) (supine) will be reported.
Number of Participants with Clinically Significant Abnormalities in Laboratory Safety Tests | Up to Week 28
  Number of participants with clinically significant abnormalities in laboratory safety tests will be reported.

SECONDARY OUTCOMES:
Change from Baseline in Villus Height to Crypt Depth (Vh:Cd) Ratio | Baseline and Week 16
  Change from baseline in Vh:Cd ratio will be reported.
Change from Baseline in Number of Intraepithelial Lymphocytes (IELs). | Baseline and Week 16
  Change from baseline in number of IELs will be reported.
Change from Baseline in Marsh-Oberhuber Scores | Baseline and Week 16
  Change from baseline in marsh-oberhuber scores will be reported. Marsh-Oberhuber score is a classification system which grades histology specimens on 6 levels from normal to total villus atrophy to characterize tissue.
Change from Baseline in Celiac Disease Symptom Diary (CDSD) Scores | Baseline and Week 16
  Change from baseline in CDSD scores will be reported. The CDSD is a daily electronic patient-reported outcome (ePRO) assessing the presence or absence of a broad range of celiac disease symptoms (diarrhea, spontaneous bowel movements, abdominal pain, bloating, nausea and tiredness). The CDSD includes 2 types of scores: a weekly symptom-specific severity score and a weekly total score. For each of the symptoms there is a possible score of 0 to 70. The total score for each week is then calculated by dividing each symptom-specific score by 10 and then summing them to get a possible total score of 0 to 70.
Change from Baseline in Celiac Disease-Gastrointestinal Symptom Rating Scale (CeD-GSRS) Score | Baseline and Week 16
  Change from baseline in CeD-GSRS will be reported. The CeD-GSRS is a modified version of the gastrointestinal symptom rating scale (GSRS). The GSRS is a questionnaire consisting of 15 symptom-specific items each graded on a 7-point Likert scale each with descriptive anchor. The scores are calculated by taking the mean of items within each of five scales: Abdominal Pain (AP), reflux, diarrhea, indigestion and constipation. The CeD-GSRS assesses 10 questions of the original GSRS. Higher scores represent more severe symptoms.
Serum Concentrations of Guselkumab | Up to Week 28
  Serum concentrations of guselkumab over time, including steady-state concentrations will be reported.
Number of Participants with Antibodies to Guselkumab | Up to Week 28
  Number of participants with antibodies to guselkumab will be reported.
Number of Participants with Neutralizing Antibodies to Guselkumab | Up to Week 28
  Number of participants with neutralizing antibodies to guselkumab will be reported.
Change from Baseline in Clinical Biomarkers High-Sensitivity C-Reactive Protein (hs-CRP) | Baseline, up to Week 28
  Change from baseline in clinical biomarker hs-CRP will be reported.
Change from Baseline in Clinical Biomarker Fecal Calprotectin | Baseline, up to Week 28
  Change from baseline in clinical biomarker fecal calprotectin will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (4):
- United States (4):
  - Clinical Trials Network, Lancaster, California
  - Clinical Research Institute of Michigan, LLC, Chesterfield, Michigan
  - West Michigan Clinical Research Center, Wyoming, Michigan
  - Hightower Clinical, Oklahoma City, Oklahoma

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency